CLINICAL TRIAL: NCT01785498
Title: Healthy Lifestyles for Children With Complex Heart Problems
Acronym: ReACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Variety Village (Unknown); Heart and Stroke Foundation of Ontario (Other); City of Toronto Parks, Forestry and Recreation (Unknown)
Responsible Party: Principal Investigator, Dr. Pat Longmuir, Scientist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB12/04X; 2012-06-1-4460033 (Other Grant/Funding Number: Ministry of Health Promotion and Sport Healthy Communities Fund)
Record Dates: First submitted 2013-02-04; First posted 2013-02-07 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Congenital Heart Defects; Inherited Cardiac Arrhythmias; Cardiomyopathy
Keywords: children; quality of life; physical activity; healthy lifestyle
MeSH Terms: conditions — Heart Defects, Congenital; Cardiomyopathies; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Receive standard clinical care and supports.
- Supplementary resources (Experimental): Receive standard care and supports plus supplementary resources developed for the intervention.
  Interventions: Behavioral: Supplementary resources

INTERVENTIONS:
Behavioral: Supplementary resources — Clinical and educational resources for patients, their families and the professionals who care for them.
  Arms: Supplementary resources

SUMMARY:
Healthy Lifestyles for Children with Complex Heart Problems is a planning and resource development project. The goal of the project is to develop an implementation plan that would enable children with complex heart problems to lead healthy, active lives within their own community. The primary goal of the project is to promote physical activity, because the physical and mental health benefits of activity are very important for these children. Children with complex heart problems have a higher risk for obesity, diabetes, acquired heart disease and mental health problems than their healthy peers. The physical health benefits of physical activity are well known, but physical activity is also key for children's mental health. Physical activity enables children to socialize with peers and create bonds and friendships. Physical activity participation also directly elevates mood through the release of brain chemicals. Children with complex heart problems are also known to experience fear and anxiety related to physical activity. This project will also develop strategies to promote healthy eating and the prevention of physical activity-related injuries to these children and their families. Children with complex heart problems are at higher risk of overweight and obesity and face unique injury risks related to pacemakers or their medications.

Extensive consultations with families and caregivers have identified needed supports for physical activity lifestyles, mental health, healthy eating and injury prevention for these children. The goal of the interviews was to understand the positive and negative influences on physical activity and healthy lifestyles for these children. Analyses of the interview content was used to develop a detailed, step-by-step implementation plan to provide the supports necessary for children with complex heart problems to lead active, healthy lives in their own community, with their family and friends. The implementation plan specifies changes to family education and counselling resources, clinical care routines, and communication among professionals and families.

The clinical trial will evaluate the impact of implementing the family supports and changes to practice previously developed. Surveys will be completed by families attending the cardiac clinic before and after the changes to practice and additional resources are made available. Interviews will be utilized to gather additional feedback from professionals and families that receive counselling utilizing the supplementary materials.

ELIGIBILITY:
Inclusion Criteria:

* child with a heart condition requiring on-going follow up between 4 and 17 years of age or parent or healthcare provider of such a child
* able to verbally answer questions and express opinions in English or French
* able to provide informed consent or assent to participate

Exclusion Criteria:

* disability other than heart condition which significantly impacts physical activity participation or healthy lifestyle habits

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Family perception of clinical service | Within 2 weeks of clinic visit
  Likert scales to measure family satisfaction with healthy lifestyle information and resources provided during clinic visit.
Pediatric Quality of Life Inventory (PedsQL) | Within 2 weeks of clinic visit

SECONDARY OUTCOMES:
Change from Baseline of Children's Self-Perceived Adequacy and Predilection for Physical Activity | 1 month after intervention completion

OTHER OUTCOMES:
Change from Baseline in Multi-dimension anxiety scale for children | 1 month after intervention completion
Change from Baseline in Pediatric Symptom Checklist | 1 month after intervention completion
Change from Baseline in PedsQL Family Impact Module | 1 month after intervention completion

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada